CLINICAL TRIAL: NCT06706570
Title: PIK3CA Mutational Status Assessment: Towards a "Tailored" Diagnostic Approach
Brief Title: PIK3CA Mutational Status Assessment
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 2029
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of PIK3CA mutational status: a route towards a tailored diagnostic approach.

DETAILED DESCRIPTION:
Evaluate the effectiveness and concordance of molecular methods in identifying mutations affecting the PIK3CA gene both on paraffin tissue sections of the tumor and on liquid biopsy of patients with breast cancer treated at the IEO. The molecular test on the liquid biopsy of same patient could bring an important benefit considering that the withdrawal of this biomaterial turns out to be less invasive than a biopsy performed on an organ

ELIGIBILITY:
Inclusion Criteria:

* • Participant has a histologically and/or cytologically confirmed diagnosis of ER+ and/or PgR+ breast cancer by local laboratory.

  * Participant has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (Fluorescent in situ hybridization (FISH), Chromogenic in situ hybridization (CISH), or Silver-enhanced in situ hybridization (SISH)) test is required by local laboratory testing.
  * Participants should be at advanced or metastatic setting prior to treatment.
  * Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.
  * Patients must be accessible for follow-up.

Exclusion Criteria:

patients already treated with different treatments like chemotherapy, hormone therapy etc

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of n=100 PIK3CA-mutant HR+/HER2- metastatic breast cancer patients will be prospectively collected. The mutational status of PIK3CA will be assessed on patients' FFPE metastasis sample tissues using a NGS panel, which covers the entire length of PIK3CA (full gene coverage). Patients with mutant PIK3CA status will be involved in the study and their FFPE as well as plasma samples will be profiled with all the different techniques (one remaining NGS panel and 2 RT-PCR assays).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of PIK3CA mutational status: a path towards a "tailored" diagnostic approach. | 2 years
  Investigate concordance between sequencing panels again generation (NGS) based on different principles and different RT-PCR assays in detecting mutations of PIK3CA.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fusco, MD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- European Institute of Oncology, Milan, MI, Italy